CLINICAL TRIAL: NCT02371031
Title: FDOPA-PET/MRI for the Pre-operative Evaluation of Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding source for study ended.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201502019
Record Dates: First submitted 2015-02-09; First posted 2015-02-25 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Glioma; Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — fluorodopa F 18; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: FDOPA-PET/MRI (Experimental): * Patients with known or suspected brain gliomas that are non-enhancing or have substantial non-enhancing regions will undergo FDOPA-PET/MRI within 2 weeks prior to planned standard of care surgical resection and/or stereotactic biopsy. In the same planning session, the MRI alone will be reviewed and then the FDOPA-PET data will be added to the planning.
  * In the event that a patient cannot undergo MRI or PET/MRI is not available (e.g. due to maintenance), FDOPA-PET/CT can be performed instead at the discretion of the responsible physician.
  * When feasible and at the discretion of the neurosurgeon performing the resection, areas of suspected tumor identified on the FDOPA-PET/MRI study but not the MRI alone will undergo tissue sampling.
  Interventions: Drug: 6-[F-18]-Fluoro-L-3,4,-dihydroxyphenylalanine; Device: PET/MRI; Procedure: Surgical resection (standard of care)

INTERVENTIONS:
Drug: 6-[F-18]-Fluoro-L-3,4,-dihydroxyphenylalanine
  Other Names: Fluorodopa; FDOPA
Device: PET/MRI
Procedure: Surgical resection (standard of care)

SUMMARY:
This is a pilot study designed to evaluate the potential of using FDOPA-PET/MRI for improving surgical planning and providing non-invasive prognostic information in patients with gliomas that have substantial non-enhancing regions. The results will be used to develop larger adequately powered studies.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected diagnosis of intracranial glioma with substantial non-enhancing regions as assessed by contrast enhanced MRI. For the purposes of this study, gliomas with substantial non-enhancing regions are defined as having contrast-enhancing volumes of less than 50% of the total estimated tumor volume. Gliomas that do not have any contrast-enhancing regions are eligible for this study.
* Standard of care surgical resection and/or stereotactic biopsy of the brain tumor planned within 2 weeks of the FDOPA-PET/MRI study.
* At least 18 years of age.
* Measurable disease on MRI defined as tumor measuring at least 1 cm in two perpendicular dimensions.
* Karnofsky performance of > 50 corresponding to ECOG categories 0, 1, or 2. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) > 30 mL/min/1.73 m^2
* Patient or legally authorized representative must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients undergoing PET/MRI: contraindication to gadolinium contrast enhanced brain MRI (i.e., allergy to gadolinium contrast, MRI-incompatible implantable devices, GFR < 30 mL/min/1.73, and severe claustrophobia). At the discretion of the responsible physician, FDOPA-PET/CT may be performed if PET/MRI is contraindicated or unavailable. If FDOPA-PET/CT is performed, the patient must have undergone a contrast-enhanced MRI for fusion with FDOPA-PET no more than 4 weeks before the FDOPA-PET/CT.
* Prior chemotherapy or radiation therapy for the brain tumor. Prior biopsy or surgical resection of the glioma without additional therapy is not an exclusion criterion.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative urine or serum pregnancy test no more than 3 days prior to FDOPA injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of cases in which the addition of FDOPA-PET to MRI changes the surgical plan | At the time of surgery (approximately week 2)
  We will consider our primary endpoint successful if FDOPA-PET changes the surgical plan in at least 4 of the 20 patients (20%), a much lower margin than previously reported with [C-11]methionine which is on the order of 60-70% of cases. When safe and feasible, these discrepant areas identified on FDOPA-PET/MRI will undergo tissue sampling. However, tissue sampling of discrepant areas may not be possible in all patients, and this decision will be made by the treating neurosurgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu